CLINICAL TRIAL: NCT03398798
Title: Analysis of Orthodontic Tooth Movement Using 3D Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-1446
Record Dates: First submitted 2017-12-15; First posted 2018-01-12 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Tooth Crowding; Dental Crowding; Malocclusion
Keywords: archwire dimension; ligation method; bracket type
MeSH Terms: conditions — Malocclusion; Crowding

STUDY DESIGN:
Intervention Model Description: There will be four different groups in this study, with each planned to consist of 20 patients (40 dental arches).
  In the twin bracket cohort, 40 dental arches are planned to be treated with .014" dimension wire, and 40 dental arches are planned to be treated with .016" dimension wire.
  In the self-ligating bracket cohort, 40 dental arches are planned to be treated with .014" dimension wire, and 40 dental arches are planned to be treated with .016" dimension wire.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Neither subjects nor the treating orthodontists will know whether a .014" or 0.16" dimension wire is being used. The investigator will assign wire dimensions using a random number generator and distribute the wires to the treating orthodontists with the archwire dimension number removed from the package. The outcomes assessor will be blinded as to which patients were treated with which archwires while analyzing the digital models of the teeth.
  Because there is a clear visual difference between twin and self-ligating brackets, there will be no blinding with regard to ligation method (bracket type).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- .014" with twin brackets (Active Comparator): .014" dimension CuNiTi orthodontic arch wires and .022" slot Ormco Insignia Metal Twin brackets.
  Interventions: Device: .014"; Device: Twin brackets
- .016" with twin brackets (Active Comparator): .016" dimension CuNiTi orthodontic arch wires and .022" slot Ormco Insignia Metal Twin brackets.
  Interventions: Device: .016"; Device: Twin brackets
- .014" with self-ligating brackets (Active Comparator): .014" dimension CuNiTi orthodontic arch wires and .022" slot Ormco Insignia SL (self-ligating) brackets.
  Interventions: Device: .014"; Device: Self-ligating brackets
- .016" with self-ligating brackets (Active Comparator): .016" dimension CuNiTi orthodontic arch wires and .022" slot Ormco Insignia SL (self-ligating) brackets.
  Interventions: Device: .016"; Device: Self-ligating brackets

INTERVENTIONS:
Device: .014" — .014" CuNiTi orthodontic arch wire
  Arms: .014" with self-ligating brackets; .014" with twin brackets
Device: .016" — .016" CuNiTi orthodontic arch wire
  Arms: .016" with self-ligating brackets; .016" with twin brackets
Device: Twin brackets — Ormco Insignia Metal Twin brackets
  Arms: .014" with twin brackets; .016" with twin brackets
Device: Self-ligating brackets — Ormco Insignia SL brackets
  Arms: .014" with self-ligating brackets; .016" with self-ligating brackets

SUMMARY:
Purpose: This project aims to study the effects of wire dimension and ligation method (bracket type) on the first stage of orthodontic treatment using 3D imaging.

Participants: Up to 80 patients at UNC School of Dentistry or Selden Orthodontics between the ages of 10 and 45, inclusive, who have been previously diagnosed with malocclusion requiring orthodontic treatment (braces) and are otherwise healthy.

Procedures (methods): Subjects receiving standard of care (SOC) orthodontic treatment will be randomized to one of two commonly used orthodontic archwires (.014" or .016" diameter). Subjects will be further subdivided for analysis based on the type of bracket (twin or self-ligating) that their clinician uses in their treatment. We will review the 3D digital images of each subject's dentition recorded as part of SOC at the 0-, 6- and 12-week visits. We will retrieve the archwires when they are removed per SOC by the clinician at the 12-week time point.

DETAILED DESCRIPTION:
Many archwire dimensions and two main bracket types (twin and self-ligating) are available to orthodontists for the first stage of orthodontic treatment, but little objective clinical evidence is available to indicate which archwire dimension and bracket type is ideal for a given patient with an individual type and degree of malalignment during this stage. A limited clinical trial will be conducted to collect and analyze this data.

The aim of this study is to study the effect of wire dimension, timing and ligation method on leveling and aligning in orthodontic treatment using 3D imaging.

The study's specific aims are as follows:

1. To analyze the effect of wire dimension (.014" vs. .016") and time-course (first six weeks or second six weeks) on Stage I treatment
2. To correlate clinical tooth movements with bench data for four types of malalignment

   1. In-out
   2. Rotation
   3. Tip
   4. Vertical step
3. To analyze the effect of ligation method (twin vs. self-ligating) on Stage I treatment

These specific aims will serve to address the following hypothesis: Archwire dimension affects tooth movement in Stage I of orthodontic treatment, depending upon variation time-course (due to force decay of superelastic wires) and method of ligation (bracket type). This will be tested in a total of 80 patients who are undergoing active treatment in the University of North Carolina (UNC) orthodontic graduate clinic or at Selden Orthodontics. There will be four different groups in this study. In the twin bracket cohort, half the patients will be treated with .014" dimension wire and half will be treated with .016" dimension wire. In the self-ligating bracket cohort, half the patients will be treated with .014" dimension wire, and half will be treated with .016" dimension wire.

If the hypotheses are shown to be correct, then the subset of society receiving orthodontic treatment will be able to benefit from selection of bracket types and archwire dimensions that match their individual types and degrees of malalignment. This will allow for more efficient tooth movement with less unwanted movement, and could lead to shorter treatment times and less discomfort.

ELIGIBILITY:
Inclusion Criteria:

* In the initial stage of active treatment at the University of North Carolina graduate orthodontic clinic or Selden Orthodontics
* Non-extraction treatment
* Maxillary and mandibular Little Index between 1-15 mm (this is a measurement of crowding)
* Presence of all permanent anterior teeth
* Age 10-45 years
* Consent to participate in the study

Exclusion Criteria:

* Systemic diseases such as diabetes, hypertension, temporomandibular disorders (TMD), craniofacial syndrome, etc.
* Any spacing between anterior teeth
* Subjects who have incisor mandibular plane angle (IMPA) greater than or equal to 100 degrees
* Anterior tooth completely blocked from the arch form
* Periodontal pocketing of any teeth greater than 4 mm
* Maxillary and mandibular Little Index >15 mm (This is a measurement of crowding. A Little Index of >15 mm indicates a need for a smaller dimension arch wire)

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chang Ko, DDS, PhD, Principal Investigator — UNC-CH
Locations (2):
- United States (2):
  - UNC-CH School of Dentistry, Chapel Hill, North Carolina
  - Selden Orthodontics, Huntersville, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- .014" With Self-ligating Brackets: .014" dimension CuNiTi orthodontic arch wires and .022" slot Ormco Insignia SL (self-ligating) brackets.
  .014": .014" CuNiTi orthodontic arch wire
  Self-ligating (SL) brackets: Ormco Insignia SL brackets
Period: Overall Study
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.2 (3.4) | 14.4 (2.2) | 14.9 (2.7) | 18.0 (6.4) | 16.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 4 | 20
  Male | 4 | 4 | 3 | 5 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Little's Index From Baseline to 6 Weeks
Description: Little's Index measures the distance between contact points on adjacent teeth. Little's Index will be measured at two time points (0 weeks and 6 weeks).
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 9 | 9 | 9 | 9
mm | -2.5 (2.2) | -2.9 (1.8) | -2.3 (1.8) | -2.6 (2.4)

2. Primary Outcome: Change in Little's Index From 6 Weeks to 12 Weeks
Description: Little's Index measures the distance between contact points on adjacent teeth. Little's Index will be measured at two time points (6 weeks and 12 weeks).
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 9 | 9 | 9 | 9
mm | -0.8 (1.0) | -0.9 (0.8) | -0.2 (0.7) | -0.4 (0.8)

3. Secondary Outcome: Linear Change in Tooth Position From Baseline to 6 Weeks (Translation)
Description: Clinical linear measurements (mm) in x-, y-, and z-translation will be measured at two time points (0 weeks and 6 weeks) to determine the linear (translational) change in tooth position during that time.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 9 | 9 | 9 | 9
mm
  Translation along the x-axis | .03 (.15) | -.05 (.18) | -.14 (.28) | -.09 (.23)
  Translation along the y-axis | .05 (.09) | .03 (.21) | -.08 (.12) | .06 (.34)
  Translation along the z-axis | -.23 (.34) | -.18 (.28) | -.22 (.3) | -.28 (.47)

4. Secondary Outcome: Linear Change in Tooth Position From 6 Weeks to 12 Weeks (Translation)
Description: Clinical linear measurements (mm) in x-, y-, and z-translation will be measured at two time points (6 weeks and 12 weeks) to determine the linear (translational) change in tooth position during that time.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 9 | 9 | 9 | 9
mm
  Translation along the x-axis | .05 (.08) | .05 (.20) | .01 (.11) | .03 (.17)
  Translation along the y-axis | .03 (.24) | .03 (.13) | -.01 (.09) | .03 (.18)
  Translation along the z-axis | -.16 (.32) | .00 (.22) | -.07 (.23) | .00 (.15)

5. Secondary Outcome: Angular Change in Tooth Position From Baseline to 6 Weeks (Rotation)
Description: Clinical angular measurements (degree) in x-, y-, and z-rotation will be measured at two time points (0 weeks and 6 weeks) to determine the angular (rotational) change in tooth position during that time.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 9 | 9 | 9 | 9
degrees
  Rotation around the x-axis | 1.95 (3.09) | 1.52 (2.84) | 1.97 (2.47) | 1.91 (3.17)
  Rotation around the y-axis | 1.37 (1.71) | .99 (1.26) | 1.33 (1.99) | 1.78 (2.50)
  Rotation around the z-axis | .66 (1.54) | .79 (1.10) | .95 (1.45) | 1.59 (3.21)

6. Secondary Outcome: Angular Change in Tooth Position From 6 Weeks to 12 Weeks (Rotation)
Description: Clinical angular measurements (degree) in x-, y-, and z-rotation will be measured at two time points (6 weeks and 12 weeks) to determine the angular (rotational) change in tooth position during that time.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 9 | 9 | 9 | 9
degrees
  Rotation around the x-axis | .82 (2.00) | 1.07 (1.81) | .66 (1.50) | .40 (1.59)
  Rotation around the y-axis | .86 (2.13) | .39 (1.34) | .40 (1.08) | -.10 (1.33)
  Rotation around the z-axis | .16 (1.33) | .18 (.83) | -.13 (1.21) | -.68 (2.21)

7. Secondary Outcome: Correlation Between Degrees of Malalignment and Rate of Tooth Movement
Description: A repeated measure linear regression model conducted to evaluate any correlation between the degrees of malalignment and the rate of tooth movement.
Time Frame: Baseline and 12 weeks
Population: Due to loss of key study personnel these data were not collected
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the study, a total 12 weeks.
Arm/Group | .014" With Twin Brackets | .016" With Twin Brackets | .014" With Self-ligating Brackets | .016" With Self-ligating Brackets
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT03398798/Prot_SAP_000.pdf